CLINICAL TRIAL: NCT06169202
Title: A Real-world Observational Study of Fruquintinib in Combination With Irinotecan and Capecitabine for the Second-line Treatment of Patients With Advanced Colorectal Cancer
Brief Title: A Study of Fruquintinib in Combination With Irinotecan and Capecitabine for the Second-line Treatment of Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Other Study IDs: FIRELIGHT
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Fruquintinib; Irinotecan; Capecitabine; Gastrointestinal Tumours
MeSH Terms: interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fruquintinib in combination with irinotecan and capecitabine: Phase I: Treatment phase: 6-8 cycles (as determined by the researcher) 1. Irinotecan: 180 mg/m2, IV, day 1, repeated every 3 weeks. (Note: If patient has UGT1A1*28 and *6 as pure or double heterozygous variants, irinotecan dose 150 mg/m2, IV, day 1, repeated every 3 weeks, with close clinical observation).
  2, Capecitabine: 1000 mg/m2 orally twice daily, D1-14, repeated every 3 weeks. 3. Fruquintinib: 4 mg orally once daily, D1-14, repeated every 3 weeks.
  Phase II: Maintenance phase:
  1, Fruquintinib: 4 mg orally once daily, D1-14, repeated every 3 weeks. 2. Capecitabine: 1000 mg/m2 orally twice daily, D1-14, repeated every 3 weeks
  Interventions: Device: fruquintinib; Drug: Irinotecan; Drug: Capecitabine

INTERVENTIONS:
Device: fruquintinib — 4 mg orally once daily, D1-14, repeated every 3 weeks.
  Other Names: elunate
Drug: Irinotecan — 180 mg/m2, IV, day 1, repeated every 3 weeks. (Note: If patient has UGT1A1*28 and *6 as pure or double heterozygous variants, irinotecan dose 150 mg/m2, IV, day 1, repeated every 3 weeks, with close clinical observation).
  Other Names: kaiputuo
Drug: Capecitabine — 1000 mg/m2 orally twice daily, D1-14, repeated every 3 weeks.
  Other Names: xiluoda

SUMMARY:
This is a real-world observational study of fruquintinib in combination with irinotecan and capecitabine for the second-line treatment of patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a real-world observational study of fruquintinib in combination with irinotecan and capecitabine for the second-line treatment of patients with advanced colorectal cancer..The purpose of the study is exploring the real-world efficacy and safety of fruquintinib in combination with irinotecan and capecitabine for the second-line treatment of patients with metastatic colorectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily enrolled in the study and signed an informed consent form, were compliant and cooperated with follow-up visits;
2. Patients with metastatic colorectal adenocarcinoma confirmed by pathology or histology;
3. Patients with second-line metastatic colorectal adenocarcinoma who have failed prior standard first-line treatment (recurrence within 6 months of the end of adjuvant chemotherapy is considered first-line treatment failure);
4. Tumor tissue testing at the primary or metastatic site allows enrollment in second-line therapy regardless of whether the KRAS, NRAS, or BRAF genes are wild-type or mutant, and regardless of microsatellite status as MSS/ pMMR or MSI-H/dMMR. For MSI-H/dMMR patients, first-line treatment was similarly allowed for enrollment if immunotherapy was used in the second line;
5. Age: 18-75 (inclusive of 18 and 75), male or female;
6. ECOG score: 0-1;
7. Expected survival ≥ 3 months;
8. At least one measurable lesion (based on RECIST 1.1 criteria);
9. Patients must undergo UGT1A1 genetic testing;
10. Major organs and bone marrow function were essentially normal (no blood components or cell growth factors had been used in the 14 days prior to enrollment):

1)Blood count: leukocytes ≥ 3.5 x 109 /L, neutrophils ≥ 1.5 x 109 /L, platelets ≥ 100 x 109 /L, hemoglobin ≥ 90 g/L; 2)International normalized ratio (INR) ≤ 1.5 x upper limit of normal (ULN) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN; 3)Liver function: total bilirubin ≤ 1.5 x ULN; ALT/AST/ALP ≤ 2.5 x ULN in the absence of liver metastases; ALT/AST/ALP ≤ 5 x ULN in the presence of liver metastases; 4)Renal function: serum creatinine ≤ 1.5 x ULN and creatinine clearance (CCr) ≥ 60 mL/min (see Appendix); 5)Normal cardiac function with left ventricular ejection fraction (LVEF ) ≥50% by 2D cardiac ultrasound; 11. Male or female patients of childbearing potential will voluntarily use an effective method of contraception, e.g., double-barrier contraception, condoms, oral or injectable contraceptives, intrauterine devices, etc., for the duration of the study and for 6 months after the last study dose. All female patients will be considered of childbearing potential unless the female patient is naturally menopausal, has undergone artificial menopause or sterilization (e.g., hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation, etc.), unless the female patient has a serum or urinalysis that shows no pregnancy within the 7 days prior to the study, and must be a non-lactating patient.

Exclusion Criteria:

1. Patients who are allergic to furaquintinib, irinotecan, and capecitabine;
2. Received anti-angiogenic small molecule TKI class (regorafenib, apatinib, lenvatinib, amlotinib, etc.) medications other than furoquinotinib prior to enrollment, etc;
3. Patients using furaquintinib and irinotecan prior to enrollment;
4. Those who have participated in a clinical trial of another antitumor drug within 4 weeks prior to enrollment or who are in the process of conducting another clinical trial;
5. Other malignancy within the past 5 years, except basal or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
6. The patient has any current disease or condition that interferes with drug absorption or the patient is unable to take furaquintinib orally;
7. Any surgical (except biopsy) or invasive treatment or manipulation within 4 weeks prior to the start of enrollment and the surgical incision has not completely healed (except for intravenous cannulation, puncture drainage, etc.);
8. There is pleural effusion, pericardial effusion, ascites, and it causes the patient to cause respiratory syndrome (≥ CTC AE grade 2 dyspnea);
9. Clinically significant electrolyte abnormalities as judged by the investigator;
10. Patients with current hypertension uncontrolled by medications were defined as patients who had hypertension and could not obtain good control with antihypertensive medication (systolic blood pressure ≥150 mmHg and diastolic blood pressure 100 mmHg);
11. Urine routine suggests urinary protein ≥3+ and the amount of urinary protein >3.5g in 24 hours; and
12. Patients with current GI disease such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors, or other conditions that may cause GI bleeding or perforation as determined by the investigator;
13. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months, vomiting blood, black stool, blood in stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or a thromboembolic event (including stroke events and/or transient ischemic attack) within 6 months;
14. Clinically significant cardiovascular disease including, but not limited to, acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; new-onset angina pectoris in the 3 months prior to enrollment; congestive heart failure New York Heart Association (NYHA) classification >2; ventricular arrhythmias requiring pharmacologic therapy;
15. Active or uncontrolled serious infection (≥ CTCAE grade 2 infection);
16. Women who are pregnant (positive pregnancy test prior to administration) or are breastfeeding;
17. Any other disease, clinically significant metabolic abnormality, physical examination abnormality, or laboratory test abnormality that, in the investigator's judgment, gives reason to suspect that the patient has a disease or condition for which the investigational drug is inappropriate (e.g., seizures requiring treatment), or that will interfere with the interpretation of the results of the study, or that puts the patient at high risk;
18. Known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection, i.e., HBV DNA positive (>1 × 104 copies/mL or >2000 IU/ml); known hepatitis C virus infection (HCV) and HCV antibody positive, or other hepatitis or cirrhosis;
19. In the judgment of the investigator, the patient has other factors that may affect the results of the study or cause this study to be forced to be terminated midway, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, concomitant family or societal factors that would affect the patient's safety;
20. Patients with brain metastases or/and carcinomatous meningitis;
21. Received radiotherapy within 4 weeks prior to enrollment and the lesion observed in this study was in the radiotherapy target area; Comorbidities requiring prolonged treatment with immunosuppressive drugs or systemic or topical corticosteroids at immunosuppressive doses (>10 mg/day of prednisone or other active hormones).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients between the ages of 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | one year
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease Control Rate (DCR) | one year
  Determined using RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No